CLINICAL TRIAL: NCT06367803
Title: Cost Analysis of Vascular Surgical Techniques: Comparing Limb Revascularisation and Amputation in Patients With CLTI at University Hospital Limerick
Brief Title: Cost Analysis of Vascular Surgical Techniques
Status: Completed | Type: Observational
Sponsor: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Fiona Leahy, Principal Investigator, University Hospital of Limerick
Other Study IDs: DVS010
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Whilst mortality rates and surgical limitations are widely known and understood for each intervention performed, the cost implications, in UHL, are not known. Therefore, it is deemed a matter of interest to understand these costs and weigh them against the mortality rates for each intervention if available.

DETAILED DESCRIPTION:
Surgical interventions for patients with CLTI include endovascular revascularisation, by-pass revascularisation and amputation.

Clinical outcomes vary greatly for each intervention. The 5-year mortality rate for major amputations i.e., below knee (BKA) and above knee (AKA), is reported to range from 30% to 70%, with AKA having the higher rate of mortality. Concomitant Type II diabetes increases these rates of mortality for both AKA and BKA.

Whilst mortality rates are widely known and understood for each intervention performed, the cost implications, in UHL, are not known. Therefore, it is deemed a matter of interest to understand these costs and weigh them against the mortality rates for each intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Cases where CLTI was treated surgically by a Vascular Consultant at UHL will be included in this analysis. That being individuals who underwent revascularisation procedures and/or lower limb amputation.
2. This analysis will look at cases from a set time frame, that being 1st March 2022 to 1st March 2023.

Exclusion Criteria:

1. Cases where CLTI was treated conservatively/without surgical intervention will not be included.
2. Surgical intervention outside of UHL.
3. Cases that occurred outside of the set timeframe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with CLTI and are under the care of a Vascular Surgeon at University Hospital Limerick
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
A comparative assessment of the cost implications of the surgical modalities used in the treatment of CLTI i.e., revascularisation and amputation. | 2 years
  A comparative assessment of the cost implications of the surgical modalities used in the treatment of CLTI i.e., revascularisation and amputation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Limerick, Limerick, Munster, Ireland

IPD SHARING:
Plan to Share IPD: Yes
This project has been written up for submission to an Irish Medical Journal